CLINICAL TRIAL: NCT00404833
Title: A Prospective Randomized Open-label Study to Compare Mycophenolate Mofetil and Corticosteroid With Conventional Immunosuppressive Treatment on Proteinuria in Idiopathic Membranous Nephropathy (MN) and Focal Segmental Glomerulosclerosis (FSGS)
Brief Title: Mycophenolate Mofetil in Membranous Nephropathy and Focal Segmental
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC1838-02; HARECCTR0500005
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Glomerulonephritis, Membranous; Glomerulosclerosis, Focal
Keywords: idiopathic membranous nephropathy or focal segmental glomerulosclerosis
MeSH Terms: conditions — Glomerulonephritis, Membranous; Glomerulosclerosis, Focal Segmental | interventions — Prednisolone; Mycophenolic Acid; Chlorambucil

INTERVENTIONS:
Drug: prednisolone and mycophenolate mofetil
Drug: prednisolone and chlorambucil

SUMMARY:
This is a prospective randomized open-label pilot study to investigate the effect of mycophenolate mofetil treatment in patients with abnormal urine protein excretion due to membranous nephropathy (MN) or focal segmental glomerulosclerosis (FSGS). The change in urine protein excretion will be the primary outcome studied. The treatment regimen comprising prednisolone and mycophenolate mofetil will be compared with prednisolone and chlorambucil in MN, and compared with prednisolone in FSGS. The study duration will be 12 months for each patient.

ELIGIBILITY:
Inclusion Criteria:

* abnormal urine protein excretion and biopsy-proven idiopathic membranous nephropathy or focal segmental glomerulosclerosis

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2003-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Proteinuria

SECONDARY OUTCOMES:
Adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Daniel TM Chan, Prof, Principal Investigator — Department of Medicine, Queen Mary Hospital
Locations (1):
- Queen Mary Hospital, Hong Kong, China

REFERENCES:
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952